CLINICAL TRIAL: NCT03329183
Title: High-dose FOLFIRI Versus Standard-dose FOLFIRI or FOLFOX-6 in Advanced Colorectal Cancer Patients With Wild-type UGT1A1*6 and *28: A Randomized, Opened, Phase II Clinical Trial
Brief Title: High-dose FOLFIRI in Advanced Colorectal Cancer Patients With Wild-type UGT1A1*6 and *28
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Zhan Wang, Associate Professor/Associate chief physician, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HFSFF
Record Dates: First submitted 2017-10-25; First posted 2017-11-01 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer
Keywords: Irinotecan; UGT1A1; Advanced Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HD-FOLFIRI (Experimental): Advanced CRC patients with Wild-type UGT1A1*6 and *28 receive high-dose FOLFIRI regimen (Irinotecan 260mg/m2 2h, leucovorin 400mg/m2, 5- fluorouracil 400mg/m2 , 5- fluorouracil 2400 mg/m2 46h, 14 days per course.)
  Interventions: Drug: Irinotecan
- SD-FOLFIRI (No Intervention): Advanced CRC patients with Wild-type UGT1A1*6 and *28 receive standard-dose FOLFIRI regimen (Irinotecan 180mg/m2 2h, leucovorin 400mg/m2, 5- fluorouracil 400mg/m2 , 5- fluorouracil 2400 mg/m2 46h, 14 days per course)
- SD-FOLFOX-6 (No Intervention): Advanced CRC patients with Wild-type UGT1A1*6 and *28 receive standard-dose FOLFOX-6 regimen (Oxaliplatin 130mg/m2 2h, leucovorin 400mg/m2, 5- fluorouracil 400mg/m2 , 5- fluorouracil 2400 mg/m2 46h, 14 days per course)

INTERVENTIONS:
Drug: Irinotecan — High-dose FOLFIRI regimen (Irinotecan 260mg/m2 2h, leucovorin 400mg/m2, 5- fluorouracil 400mg/m2 , 5- fluorouracil 2400 mg/m2 46h, 14 days per course)
  Other Names: CPT-11
  Arms: HD-FOLFIRI

SUMMARY:
This trial aims to evaluate the efficacy, safety of high-dose FOLFIRI regimen in advanced colorectal cancer patients with wild-type UGT1A1*6 and *28.

DETAILED DESCRIPTION:
Pharmacogenetic testing of uridine diphosphate glucuronosyltransferase 1A1 (UGT1A1) *6/*28 is recommended in clinical practice prior to the administration of irinotecan (CPT-11)-based regimens, such as FOLFIRI regimen in patients with advanced colorectal cancer. To avoid severe toxicity of irinotecan, such as severe neutropenia and diarrhea, patients with UGT1A1 *6/*28 mutation often start with a reduced dose of irinotecan. However, it remains unclear whether high-dose CPT-based regimen (FOLFIRI) could increase clinical efficacy in CRC patients when compared with standard-dose FOLFIRI or FOLFOX-6 regimens. This trial aims to compare the efficacy, safety of high-dose FOLFIRI and standard-dose FOLFIRI or FOLFOX-6 in advanced colorectal cancer patients with UGT1A1*6 G/G and *28 TA6/6.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be histologically diagnosed with advanced colorectal adenocarcinoma or postoperative recurrence
* Patients should be with UGT1A1*28 wild-type TA6/6 and UGT1A1*6 wild-type G/G
* Patients have measurable lesions
* Patients are not available for targeted therapy or patients refuse to receive targeted therapy
* Age should be more than 18 years
* Performance status should be 0-2
* Hemoglobin should be more than 9.0 g/dL; Absolute Neutrophil Count should be more than 1,500/mm3; Platelet should be more than 80,000/mm3；Total Bilirubin should be less than 1.5 times of the upper limit of normal value; Alanine aminotransferase and Glutamic-oxaloacetic transaminase should less than 2.5 times of the upper limit of normal value (it can be 5 times if liver metastasis); Creatinine should be be less than 1.5 times of the upper limit of normal value

Exclusion Criteria:

* Patients with UGT1A1*28 wild-type TA6/7, TA7/7 and UGT1A1*6 wild-type G/A,A/A;
* Patients with brain metastases;
* Patients could not tolerate chemotherapy;
* Patients have secondary primary tumor;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | up to 55 months
  Evaluation of tumor burden based on RECIST criteria every 4 cycles(each cycle is 14 days), ORR is the proportion of patients with reduction in tumor burden of a predefined amount, including complete response and partial response.

SECONDARY OUTCOMES:
Early tumor shrinkage (ETS) rate | up to 55 months
  (ETS) rate is defined as 20% reduction in target lesions after the first 6 weeks of treatment (first tumor assessment)
Disease Control Rate (DCR) | up to 55 months
  Evaluation of tumor burden based on RECIST criteria every 4 cycles(each cycle is 14 days), and DCR is the proportion of patients with reduction in tumor burden of a predefined amount, including complete response, partial response and stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Sheng Zang, Prof, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China